CLINICAL TRIAL: NCT02119091
Title: A Double-center, Randomized, Double-blinded, 2-way Crossover, Placebo-controlled Study: Comparison of Single Oral Dose 400mg Moxifloxacin-induced QT Prolongation Between Healthy Chinese Volunteers and Caucasian Volunteers
Brief Title: Race Difference Moxifloxacin-induced QT Prolongation Between Healthy Chinese and Caucasian Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haiyan Li (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); Spaulding Clinical Research LLC (Other); BioClinica, Inc. (Industry); Peking University (Other)
Responsible Party: Sponsor-Investigator, Haiyan Li, Director, Clinical Trial Center, Peking University Third Hospital, China, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PUTH_CTC_2013_001
Record Dates: First submitted 2014-04-15; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Cardiac Toxicity
Keywords: QT prolongation; Chinese; Caucasian; Moxifloxacin
MeSH Terms: conditions — Cardiotoxicity; Long QT Syndrome | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxifloxacin (Experimental): Single oral dose 400 mg
  Interventions: Drug: Moxifloxacin
- Placebo (Placebo Comparator): Single oral dose

INTERVENTIONS:
Drug: Moxifloxacin
  Arms: Moxifloxacin

SUMMARY:
A double-center, randomized, double-blinded, 2-way crossover, placebo-controlled Study: Comparison of single oral dose 400mg Moxifloxacin-induced QT prolongation between healthy Chinese volunteers and Caucasian Volunteers Study Objective:Primary Objective:To compare the difference of ΔΔQTcF (Baseline-adjusted, placebo-corrected effect on QTcF) between Chinese group and Caucasian group under the same exposure (Cmax) of Moxifloxacin.Secondary Objectives:1)To compare the difference of ΔΔQTcF, heart rate, PR, RR, QRS and Moxifloxacin plasma concentration between Chinese group and Caucasian group.2)To compare slopes of Moxifloxacin plasma Concentration/QTcF value between healthy Chinese volunteers and Caucasian Volunteers.

DETAILED DESCRIPTION:
A total 80 healthy subjects will be enrolled in both sites, both male and female, age 18-45 years old. Half of them will be healthy Chinese volunteers, both male and female; will be recruited to obtain at least 36 evaluable volunteers in Chinese site of CTC, PUTH. The other half will be healthy Caucasian volunteers, both male and female; will be recruited to obtain at least 36 evaluable volunteers in the U.S. site of Spaulding Clinical Research LLC. An evaluable subject is defined as a volunteer completing all study procedures from the screening period to the final ECG nominal time-point for QTc interval measurement and final blood sampling for plasma levels of Moxifloxacin on the last study day (Day 2 of the second period).

Study Objective:Primary Objective:To compare the difference of ΔΔQTcF (Baseline-adjusted, placebo-corrected effect on QTcF) between Chinese group and Caucasian group under the same exposure (Cmax) of Moxifloxacin.Secondary Objectives:1)To compare the difference of ΔΔQTcF, heart rate, PR, RR, QRS and Moxifloxacin plasma concentration between Chinese group and Caucasian group.2)To compare slopes of Moxifloxacin plasma Concentration/QTcF value between healthy Chinese volunteers and Caucasian Volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese subjects, male and female, 18 to 45 years of age, inclusive, and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.(only for PUTH site) Or, healthy non-Hispanic Caucasian subjects, male and female, 18 to 45 years of age, inclusive, and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening (only for SCR site).
2. At Screening and baseline day, vital signs (systolic and diastolic blood pressure and heart rate rate) will be assessed in the sitting position after the subject has rested for 5 minutes. All of vital signs should be within normal ranges:

   * Body temperature (Oral) between 35.0-37.0°C
   * 90 mm Hg ≤ systolic blood pressure <150 mm Hg
   * 50 mm Hg≤ diastolic blood pressure < 90 mm Hg
   * 50beats per minute≤ Heart rate ≤ 90 beats per minute
3. Body weight need to be at least 50kg or above, 18Kg/m2≤ Body Mass Index(BMI) ≤31Kg/m2
4. Be able to communicate well with the investigator, to understand and comply with the requirements of the study. Understand and sign the written informed consent forms prior to any screening procedures.

Exclusion Criteria:

1. Subject has a 12 lead ECG result at Screening or Check in with evidence of any of the following abnormalities after the subject has rested for approximately10 minutes.

   * QTcF>450 ms for males and females
   * PR interval >240 ms or <110 ms
   * Second-degree or third-degree atrioventricular block(AVB)
   * Complete left or right bundle branch block or incomplete left bundle branch block
   * QRS duration >120 ms
   * Heart rate <50 beats per minute or >90 beats per minute
   * Pathological Q-waves (defined as Q-wave ≥40 ms)
   * Ventricular pre-excitation
2. Subject has a history of unexplained syncope, structural heart disease, long QT syndrome, heart failure, myocardial infarction, angina, unexplained cardiac arrhythmia, torsades de points, or ventricular tachycardia. Subjects will also be excluded if there is a family history of long QT syndrome (genetically proven or suggested by sudden death of a close relative due to cardiac causes at a young age) or Brugada syndrome.
3. Subject has hypokalemia, hypocalcemia, or hypomagnesemia according to lower limits of the reference ranges provided by the clinical laboratory.
4. Subject has a history or current evidence of anaphylactic reactions or clinically significant (as determined by the investigator) allergic conditions (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
5. Subject has a hypersensitivity or allergy to moxifloxacin or any drug in the fluoroquinolone class (eg, ciprofloxacin or levofloxacin).
6. History or clinical manifestations of significant metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, urological, neurological, genetic or psychiatric disorders.
7. Current or recent history (< 30 days prior to Screening) of a clinically significant illness.
8. Use of any prescription drugs, herbal supplements, within 4 weeks prior to initial dosing, and/or over-the-counter (OTC) medication, dietary supplements (vitamins included) within 4 week prior to initial dosing.
9. Positive results of human immunodeficiency virus, Hepatitis B surface antigen or Hepatitis C antibody testing.
10. Current use of tobacco (> 10 tobacco/day) or nicotine-containing products. .
11. History of drug or alcohol abuse within the 12 months prior to dosing, or evidence of such abuse as indicated by the laboratory assays conducted during the screening and/or at baseline.
12. Dosing of study drug in any clinical investigation within 30 days prior to initial dosing.
13. Donation or loss of 200 ml or more of blood within 30 days prior to participation, or donation of component blood within 30 days prior to participation.
14. Consumption of alcohol-, caffeine -containing foods or beverages within 48 hours preceding study drug administration.
15. Females are currently pregnant, breast-feeding or planning a pregnancy in the next 3 months.
16. Other conditions which investigator deems potential harm to subjects if participate the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
ΔΔQTcF | 2 months
  To compare the difference of ΔΔQTcF (Baseline-adjusted, placebo-corrected effect on QTcF) between Chinese group and Caucasian group under the same exposure (Cmax) of Moxifloxacin

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Li, MD, Principal Investigator — Director of Clinical Trial Center,Peking University Third Hospital
Locations (2):
- Spaulding Clinical Research LLC, West Bend, Wisconsin, United States
- Peking University Third Hospital Clinical Trial Center, Beijing, Beijing Municipality, China